CLINICAL TRIAL: NCT06078514
Title: Sexual Function and Quality of Life After LEEP: a Prospective Multi-Center Study
Acronym: SEQUEL
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Hyvinkää Hospital (Other); North Karelia Central Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Laura Kotaniemi-Talonen, Deputy Chief, Gynecology and Obstetrics, Tampere University Hospital
Other Study IDs: R22017
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cervical Dysplasia
Keywords: Colposcopy; LEEP; Cervical dysplasia; HSIL; Sexual function index; Health-related quality of life
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Loop electrosurgical excision procedure (LEEP): Women directed to colposcopy examination due to cytological abnormality or repeated HPV-positivity and undergone a LEEP procedure due to HPV-related cervical lesion
  Interventions: Procedure: Loop electrosurgical excision procedure (LEEP)
- Colposcopy only: Women directed to colposcopy examination due to cytological abnormality or repeated HPV-positivity with no indication to LEEP

INTERVENTIONS:
Procedure: Loop electrosurgical excision procedure (LEEP) — The affected area of cervix is excised under local anesthesia using a small thin electrically charged hardwire loop for simultaneous cutting and electrocoagulation.
  Other Names: Large loop excision of the transformation zone (LLETZ)
  Groups: Loop electrosurgical excision procedure (LEEP)

SUMMARY:
The goal of this prospective study is to investigate the sexual function and quality of life of women undergoing loop electrosurgical excision procedure (LEEP) due to HPV-related cervical lesion.

The main question it aims to answer are:

* Whether LEEP affects the sexual function of women in comparison to untreated women, and
* Whether LEEP affects the health-related quality of life of women in comparison to untreated women

Participants are asked to complete web based an international validated self-report questionnaire on sexual function issues, the Female Sexual Function Index (FSFI), and a validated quality of life -questionnaire 15D at the time of first colposcopy appointment and six and 24 months, 3 years and 5 years after index visit (LEEP or first colposcopy in control group). Relevant additional background information is also collected via questionnaire and from patient files.

Researchers will compare women with LEEP and those with only colposcopy visits to see any differences between self-reported sexual function (FSFI scores) or health-related quality of life (15D scores) both short and long-term.

DETAILED DESCRIPTION:
We plan to recruit minimum of 1000 women referred to colposcopy in Tampere University Hospital, Helsinki University Hospital, Kuopio University Hospital, Oulu University Hospital, North Karelia Central Hospital and Hyvinkää Hospital to our prospective multi-center study. Recruitment is done at gynecology outpatient clinics of the participating units at the first colposcopy visit, where the doctor performing the colposcopy informs the eligible women about the study, gives them the patient information letter, and asks them to participate and, if they agree, to fill in the informed consent. We aim to recruit 500 women undergoing LEEP (intervention arm) and at least 500 undergoing only colposcopy (control arm).

Pirkanmaa Hospital District Ethical Review Board has approved the study design and local scientific committees in each university hospital area applied for permission to launch the study.

In each participating unit, eligible women will be given a written patient information sheet on the study and asked to participate. From women willing to participate, a written informed consent will be collected and stored in locked cabinet in participating unit. These documents will be accessed only by study members.

Participants are contacted due to the study 5 times: at the time of recruitment, 6 months after the index visit (either first colposcopy or LEEP visit) and 24 months, 3 years and 5 years after the index visit. Each time they are asked to fill in the same questionnaires, sent by mail and available also web based. No additional visits are needed, nor any extra samples taken.

The study data is collected using REDCap system designed for safe patient data management. Access to the system is strictly restricted to the research team members, that are committed to handle the data according to good clinical practice.

At the end of the study, the digital data is to be stored at Pirkanmaa Hospital Disctrict official research files, where individual patient data will be available only for identified study members. In the analysis the data will be used pseudonymized. Informed consents will be stored in participating research units.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* First colposcopy visit (in 24 months, if previous colposcopies)
* Referral for cytological changes or repeated HPV positivity
* No previous LEEP or other operations affecting the length of cervix
* Not pregnant at the time of colposcopy/LEEP
* Sexually active
* Capable of understanding the study protocol - informed consent given
* Fluent in Finnish

Exclusion Criteria:

* Age less than 18 or more than 70 years
* Previous colposcopy within 24 months
* Referral for other reason, e.g. vulvar lesion
* Previous LEEP or other operation affecting the length of cervix
* Pregnant at the time of colposcopy/LEEP
* Sexually inactive
* Unable to understand the study protocol - no informed consent
* Difficulties in understanding Finnish

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female by birth
Study Population: The study population consists of adult, sexually active, non-pregnant, 18-70 year-old women referred to gynecology outpatient clinics of the participating units for colposcopy due to cytological changes or repeated HPV positivity.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported sexual function measured by Female Sexual Function Index (FSFI) | From 6 months up to 5 years since the initiation of the study
  Female Sexual Function Index (FSFI) is a 19-item self-report measure that provides scores on overall levels of sexual function as well as the primary components of sexual function in women, including sexual desire, arousal, orgasm, pain, and satisfaction. For scoring it uses a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning on the respective item. Total that scores of ≤26.55 are considered to present clinically relevant sexual dysfunction (specificity = 0.733; sensitivity = 0.889).
Self-reported health-related quality of life measured by 15D | From 6 months up to 5 years since the initiation of the study
  15D is a generic, comprehensive, 15-dimensional, standardized, self-administered measure of health-related quality of life (HRQoL). It includes the following 15 dimensions: breathing, mental function, speech (communication), vision, mobility, usual activities, vitality, hearing, eating, elimination, sleeping, distress, discomfort and symptoms, sexual activity, and depression. The maximum score is 1 (no problems on any dimension) and the minimum score is 0. A change of 0.02-0.03 has been observed to be such that people can feel the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kotaniemi-Talonen, PhD, Principal Investigator — Tampere University Hospital
Locations (5):
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No